CLINICAL TRIAL: NCT00382187
Title: A Phase II, Randomized, Controlled, Observer-blind, Single-Center Study to Evaluate Safety and Immunogenicity of Two Doses, Administered Three Weeks Apart, and a Six Month Booster Dose of Two Surface Antigen Adjuvanted With MF59C.1 Influenza Vaccines Containing 7.5 Micrograms or 15 Micrograms of A/H5N1 Influenza Antigen and of a Non-adjuvanted Influenza Vaccine Containing 15 Micrograms of A/H5N1 Influenza Antigen, in Adults
Brief Title: Safety and Immunogenicity of Two Adjuvanted and One Non-adjuvanted H5N1 Influenza Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V87P2; Eudract number 2006-004063-66
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-02

CONDITIONS: Influenza
Keywords: influenza; pandemic influenza; influenza vaccine; adjuvanted influenza vaccine; H5N1 influenza antigen; MF59; Pandemic influenza disease
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- MF59 adjuvant H5N1 influenza vaccine 7.5 micrograms (Experimental)
  Interventions: Biological: MF59 adjuvanted H5N1 influenza vaccine
- MF59 adjuvant H5N1 influenza vaccine 15 micrograms (Experimental)
  Interventions: Biological: MF59 adjuvanted H5N1 influenza vaccine
- non-adjuvanted influenza vaccine 15 micrograms of H5N1 antigen (Experimental)
  Interventions: Biological: MF59 adjuvanted H5N1 influenza vaccine

INTERVENTIONS:
Biological: MF59 adjuvanted H5N1 influenza vaccine — * MF59 adjuvanted (H5N1) influenza vaccine (Vietnam strain) containing 7.5 mg or 15 mg of H5N1
  * non-adjuvanted influenza vaccine containing 15 ug of H5N1

SUMMARY:
The present study aims to evaluate safety and immunogenicity of two doses, administered three weeks apart, and a 6 month booster dose, of two influenza vaccines containing 7.5 micrograms or 15 micrograms of H5N1 influenza antigen, and of a non-adjuvanted influenza vaccine containing 15 micrograms of H5N1 influenza antigen, in adults

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers 18-60 years of age

Exclusion Criteria:

* Any auto-immune disease or other serious acute, chronic or progressive disease
* Hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine
* Within the past 7 days, they have experienced any acute disease or infections requiring systemic antibiotic or antiviral therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
CPMP criteria for evaluation of flu vaccines e.g. Seroprotection, GMT's and Seroconversion rate at day 0 and day 22 and day 43 following vaccination. | day 1 to day 43

SECONDARY OUTCOMES:
Solicited Local and Systemic Reactions Within 6 Days Following Each Vaccination And Adverse Events Throughout the Study. | Day 1 to Day 382

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Information Services, Study Chair — Novartis
Locations (1):
- Presidio Distrettuale N. 8, Azienda USL 7 di Siena, Via Savina Petrilli, 3, Siena, Siena, Italy

REFERENCES:
- [Result] Galli G, Medini D, Borgogni E, Zedda L, Bardelli M, Malzone C, Nuti S, Tavarini S, Sammicheli C, Hilbert AK, Brauer V, Banzhoff A, Rappuoli R, Del Giudice G, Castellino F. Adjuvanted H5N1 vaccine induces early CD4+ T cell response that predicts long-term persistence of protective antibody levels. Proc Natl Acad Sci U S A. 2009 Mar 10;106(10):3877-82. doi: 10.1073/pnas.0813390106. Epub 2009 Feb 23. PMID 19237568